CLINICAL TRIAL: NCT05096741
Title: OCS Liver PROTECT Continuation Post-Approval Study
Status: Completed | Type: Observational
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Other Study IDs: OCS-LVR-01-PAS
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Liver Transplant

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- OCS Liver
  Interventions: Device: OCS Liver
- Control

INTERVENTIONS:
Device: OCS Liver — Transplanted with a OCS preserved liver
  Groups: OCS Liver

SUMMARY:
Post-approval observational study of subjects that were enrolled and transplanted in the OCS Liver PROTECT Trial.

DETAILED DESCRIPTION:
Post-approval observational study of subjects that were enrolled and transplanted in the OCS Liver PROTECT Trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects transplanted in the OCS Liver PROTECT Trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects transplanted in the OCS Liver PROTECT Trial
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-01-24 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Liver Graft Survival | 2 years
  Liver Graft Survival through 2 years (24 months) after transplantation.

OTHER OUTCOMES:
Patient Survival | 2 years
  Patient Survival (freedom from mortality) through 2 years (24 months) after transplantation.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - University of California San Diego, La Jolla, California
  - Scripps, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Tampa General, Tampa, Florida
  - Emory, Atlanta, Georgia
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - University of Texas Southwest, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - University of Washington, Seattle, Washington